CLINICAL TRIAL: NCT01973686
Title: Active Commuting To Improve Well-being and Health in Everyday Life (ACTIWE)
Brief Title: GO-ACTIWE Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bente Merete Stallknecht, Professor, University of Copenhagen
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ACTIWE-2
Record Dates: First submitted 2013-10-21; First posted 2013-10-31 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vigorous intensity LTPA (Experimental): Leisure time physical activity (LTPA): Exercise intensity: 70% of maximal oxygen uptake (VO2 max); Energy expenditure: Females: 1600 kcal/week; Males: 2100 kcal/week
  Interventions: Behavioral: Physical activity
- Moderate intensity LTPA (Experimental): Leisure time physical activity (LTPA): Exercise intensity: 50% VO2 max; Energy expenditure: Females: 1600 kcal/week; Males: 2100 kcal/week
  Interventions: Behavioral: Physical activity
- Control (No Intervention): Receives no intervention

INTERVENTIONS:
Behavioral: Physical activity
  Arms: Moderate intensity LTPA; Vigorous intensity LTPA

SUMMARY:
The aim of the present study is to investigate the changes in body composition and the degree of compensation to exercise induced energy expenditure after 1 year of physical activity with either moderate or vigorous intensity in overweight and class 1 obese men and women. The present study is a sub study to main study "Active Commuting To Improve Well-being and Health in Everyday Life" (NCT 01962259)

ELIGIBILITY:
Inclusion Criteria:

* Participation in main study (NCT 01962259)

Exclusion Criteria:

* No participation in main study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Total body fat | Change from baseline in body fat at 3 months
  Changes in total body fat (kg) measured by dual x-ray absorptiometry
Total body fat | Change from baseline in body fat at 6 months
  Changes in total body fat (kg) measured by dual x-ray absorptiometry

SECONDARY OUTCOMES:
Net energy balance and degree of compensation | 3 and 6 months
  1. Net energy balance calculated from changes in body composition, and 2. the degree of compensation as the difference between energy spent during exercise and net energy balance
Compensatory mechanisms | Baseline, 3 and 6 months
  1. Resting metabolic rate determined by indirect calorimetry, 2. Total physical activity (TPA) measured using accelerometry, 3. Non-exercise activity determined as the difference between TPA and exercise activity, and 4. Energy intake determined by food records and during meal tests
Appetite control | Baseline, 3 and 6 months
  Appetite control determined via 1. blood samples (peptides and metabolites) and 2. self rated sensations (visual analogue scales) in relation with standardized meals and exercise, as well as 3. ad libitum energy intake and 4. Eating behaviours determined via three-factor eating questionaire
Anthropometry | Baseline, 3 and 6 months
  Body composition measured by dual x-ray absorptiometry, height, weight, waist and hip circumference, sagittal abdominal height

OTHER OUTCOMES:
Exercise compliance and energy expenditure | Baseline, 3 and 6 month
  Exercise compliance and energy expenditure will be measured and adjusted continuously with the use of heart rate monitors over the course of the 1 year intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bente M Stallknecht, MD PhD DMSc, Principal Investigator — Professor
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen, Denmark

REFERENCES:
- [Derived] Quist JS, Rosenkilde M, Petersen MB, Gram AS, Sjodin A, Stallknecht B. Effects of active commuting and leisure-time exercise on fat loss in women and men with overweight and obesity: a randomized controlled trial. Int J Obes (Lond). 2018 Mar;42(3):469-478. doi: 10.1038/ijo.2017.253. Epub 2017 Oct 10. PMID 28993707